CLINICAL TRIAL: NCT03092934
Title: A Phase I/II Open-Label Multicenter Study to Evaluate the Safety and Efficacy of AK-01 as Monotherapy in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of AK-01 (LY3295668) in Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: AurKa Pharma Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17228; AURA-001 (Other: AurKa Pharma Inc.); J1O-MC-JZHA (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Results first posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Neoplasms; Neoplasm Metastasis; Triple Negative Breast Neoplasms; Head and Neck Neoplasms; Breast Neoplasms; Solid Tumor, Adult; Small Cell Lung Carcinoma
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Triple Negative Breast Neoplasms; Head and Neck Neoplasms; Breast Neoplasms; Small Cell Lung Carcinoma | interventions — LY3295668 erbumine

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 25 milligrams (mg) LY3295668 (Phase 1) (Experimental): 25 milligrams (mg) LY3295668 twice daily (BID) administered orally in 21-day cycles.
  Interventions: Drug: LY3295668
- 50 mg LY3295668 (Phase 1) (Experimental): 50 mg LY3295668 BID administered orally in 21-day cycles.
  Interventions: Drug: LY3295668
- 75 mg LY3295668 (Phase 1) (Experimental): 75 mg LY3295668 BID administered orally in 21-day cycles.
  Interventions: Drug: LY3295668
- 25 mg LY3295668 (Phase 2) (Experimental): 25 mg LY3295668 BID administered orally in 21-day cycles.
  Interventions: Drug: LY3295668

INTERVENTIONS:
Drug: LY3295668 — Oral capsules
  Other Names: AK-01; Erbumine

SUMMARY:
This two-part study consists of a phase 1 dose escalation study in participants with locally advanced or metastatic solid tumors, and a phase 2 portion in up to 3 groups with either small cell lung cancer, breast cancer and/or one other solid tumor type.

ELIGIBILITY:
Inclusion Criteria:

* Have received at least 1 but no more than 4 prior systemic therapies
* Have adequate organ function
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have estimated life expectancy greater than or equal to (≥)12 weeks
* Have fully recovered from radiation therapy or surgery, and are recovering from any acute adverse effects of other cancer therapies
* Have discontinued all chemotherapy, investigational therapy, molecularly-targeted therapy, and cancer-related hormonal therapy at least 14 days prior, biologic or immunotherapeutic therapy at least 21 days prior, or mitomycin-C or nitrosoureas at least 6 weeks prior
* Female participants with reproductive potential agree to use 2 forms of highly effective contraception during the study and for the following 3 months
* Male participants must use a barrier method of contraception during the study and for the following 3 months

Phase 1

* Have evidence of a solid tumor that is locally advanced and/or metastatic (excluding primary brain tumor)

Phase 2

* Have disease measurable by Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1
* Have evidence of a solid tumor that is locally advanced and/or metastatic, and in:

  * Small Cell Lung Cancer (SCLC), must have failed platinum-containing therapy
  * Breast Cancer, be Estrogen Receptor positive and/or Progesterone Receptor positive, but Human Epidermal Growth Factor Receptor 2 (HER2) negative, and must have failed a hormone therapy and a Cyclin-dependent kinase 4/6 (CDK4/6) inhibitor
  * Triple negative breast cancer (TNBC) and failed standard therapy
  * Squamous cell cancers of the head neck associated with the human papilloma virus (HPV), and have failed standard therapy
  * Other solid tumor type that has been approved by the sponsor

Exclusion Criteria:

* Have symptomatic central nervous system (CNS) metastasis (unless asymptomatic and not current receiving corticosteroids) or a primary tumor of the CNS
* Have a medical condition that precludes participation (swallowing disorder, organ transplant, pregnant or nursing, HIV, active Hepatitis B or C, cardiac disease, history of major surgery in upper gastrointestinal (GI) tract or GI disease, hypokalemia, hypomagnesaemia or hypocalcaemia that cannot be controlled)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Jewish General Hospital, Montreal, Quebec
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Chu QS, Bouganim N, Fortier C, Zaknoen S, Stille JR, Kremer JD, Yuen E, Hui YH, de la Pena A, Lithio A, Smith PS, Batist G. Aurora kinase A inhibitor, LY3295668 erbumine: a phase 1 monotherapy safety study in patients with locally advanced or metastatic solid tumors. Invest New Drugs. 2021 Aug;39(4):1001-1010. doi: 10.1007/s10637-020-01049-3. Epub 2021 Jan 22. PMID 33479856

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase I participants are said to have completed the study if they completed Dose Limiting Toxicity (DLT) period or have had a DLT. Phase II participants who died or are alive and on study at conclusion but off treatment are defined as completed.
Groups:
- 25 Milligrams (mg) LY3295668 (Phase 1): 25 mg LY3295668 twice daily (BID) administered orally in 21-day cycles.
Period: Overall Study
Arm/Group | 25 Milligrams (mg) LY3295668 (Phase 1) | 50 mg LY3295668 (Phase 1) | 75 mg LY3295668 (Phase 1) | 25 mg LY3295668 (Phase 2)
Started | 8 | 2 | 2 | 1
Received at Least One Dose of Study Drug | 8 | 2 | 2 | 1
Completed | 8 | 2 | 2 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- 50 mg LY3295668 (Phase 1): 50 milligrams (mg) LY3295668 BID administered orally in 21-day cycles.
  LY3295668: Oral capsules
- Total: Total of all reporting groups
Arm/Group | 25 Milligrams (mg) LY3295668 (Phase 1) | 50 mg LY3295668 (Phase 1) | 75 mg LY3295668 (Phase 1) | 25 mg LY3295668 (Phase 2) | Total
Number analyzed (Participants) | 8 | 2 | 2 | 1 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 0 | 0 | 0 | 7
  >=65 years | 1 | 2 | 2 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 1 | 8
  Male | 4 | 1 | 0 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 2 | 2 | 1 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 2 | 2 | 1 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 8 | 2 | 2 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose
Description: Maximum Tolerated Dose (MTD) was defined as the dose immediately below the dose at which ≥2/3, ≥2/6, or ≥3/9 participants in a cohort experienced a dose limiting toxicity (DLT) during the first 21 days of treatment (Cycle 1) in Phase 1.
Time Frame: Cycle 1 (21 days)
Population: All participants who received at least one dose of study drug and experienced a DLT; or received ≥ 38 doses of study drug in Cycle 1 and were not discontinued from the study before completing Cycle 1.
Measure: Number; unit: milligram (mg)
Groups:
- LY3295668 Phase 1: 25 milligrams (mg) LY3295668 twice daily (BID) administered orally in 21-day cycles.
Arm/Group | LY3295668 Phase 1
Number analyzed (Participants) | 12
milligram (mg) | 25

2. Primary Outcome: Phase 2: Percentage of Participants Who Achieved Partial Response (PR) or Complete Response (CR) [Objective Response Rate (ORR)]
Description: Objective response rate (ORR) was defined as a percentage of responders who achieved complete response or partial response (CR+PR) as assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v 1.1). Complete response (CR) is defined as disappearance of all target (and non-target) lesions, and no appearance of new lesion. Partial response (PR) was defined as at least a 30% decrease in the sum of longest diameters (LD) of target lesions, taking as reference the baseline sum of LD, no progression of non-target lesions, and no appearance of new lesions.
Time Frame: Baseline to Objective Disease Progression (Up to 11 months)
Population: All patients who received at least 1 dose of AK-01, whether or not they completed all protocol requirements.
Measure: Number; unit: percentage of participants
Arm/Group | 25 mg LY3295668 (Phase 2)
Number analyzed (Participants) | 1
percentage of participants | 0

3. Secondary Outcome: Phase 1: Number of Participants With One or More Treatment-Emergent Adverse Events
Description: A treatment-emergent adverse event (AE) is an AE that started or worsened (increased in severity) from the treatment start date to 30 days after the treatment end date. A summary of other non-serious Adverse Events (AEs), and all Serious Adverse Events (SAE's), regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Cycle 1 Day 1 through 30 Days After Treatment End Date (Up to 29 Months)
Population: All participants who received at least one dose of study drug, whether or not they completed all protocol requirements.
Measure: Count of Participants; unit: Participants
Groups:
- 25 mg LY3295668 (Phase 1): 25 mg LY3295668 BID administered orally in 21-day cycles.
Arm/Group | 25 mg LY3295668 (Phase 1) | 50 mg LY3295668 (Phase 1) | 75 mg LY3295668 (Phase 1)
Number analyzed (Participants) | 8 | 2 | 2
Participants | 7 | 2 | 2

4. Secondary Outcome: Phase 2: Number of Participants With One or More Treatment-Emergent Adverse Events
Description: as for outcome 3
Time Frame: Cycle 1 Day 1 through 30 Days After Treatment End Date (Up to 29 Months)
Population: All participants who received at least one dose of study drug whether or not they completed all protocol requirements.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg LY3295668 (Phase 2)
Number analyzed (Participants) | 1
Participants | 1

5. Secondary Outcome: Phase 2: Pharmacokinetic (PK): Area Under the Plasma Concentration-time Curve From Time Zero to 12 Hours Post-dose (AUC[0-12]) (Phase 2)
Description: Area under the plasma concentration-time curve for LY3295668 from time zero to 12 hours.
Time Frame: Cycle 1: Day 1 and Day 15: Predose, 1, 2, 4, 6, and 8 - 12 hours postdose; Cycle 1: Day 2 and Day 8 predose
Population: Zero participants analyzed due to data not collected.
Arm/Group | 25 mg LY3295668 (Phase 2)
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 2: PK: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours Post-dose (AUC[0-24])
Description: Area under the plasma concentration-time curve for LY3295668 from time zero to 24 hours.
Time Frame: Cycle 1: Day 1 and Day 15: Predose, 1, 2, 4, 6, and 8-12 hours post-dose; Cycle 1: Day 2 and Day 8 Predose
Population: Zero participants analyzed due to data not collected.
Arm/Group | 25 mg LY3295668 (Phase 2)
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase 2: PK: Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration for LY3295668.
Time Frame: Cycle 1: Day 1 and Day 15: Predose, 1, 2, 4, 6, and 8 hours post-dose
Population: All participants who received at least one dose of study drug and had evaluable PK data in Phase 2 per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per liter (µg/L)
Arm/Group | 25 mg LY3295668 (Phase 2)
Number analyzed (Participants) | 1
micrograms per liter (µg/L)
  Day 1 | NA (NA) — N=1, Geometric mean and Geometric Coefficient of Variation were not calculated. Individual value reported: 4409.45 µg/L
  Day 15 | NA (NA) — N=1, Geometric mean and Geometric Coefficient of Variation were not calculated. Individual value reported: 11070.42 µg/L

8. Secondary Outcome: Phase 2: PK: Time of Maximum Observed Plasma Concentration (Tmax)
Description: Time of maximum observed plasma concentration of LY3295668.
Time Frame: Cycle 1: Day 1 and Day 15: Predose, 1, 2, 4, 6, and 8 hours post-dose
Population: All participants who received at least one dose of study drug and had evaluable PK data in Phase 2 per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | 25 mg LY3295668 (Phase 2)
Number analyzed (Participants) | 1
hours
  Day 1 | NA (NA) — N=1, Geometric mean and Geometric Coefficient of Variation were not calculated. Individual value reported: 2.03 hours.
  Day 15 | NA (NA) — N=1, Geometric mean and Geometric Coefficient of Variation were not calculated. Individual value reported: 1.03 hours.

9. Secondary Outcome: Phase 2: PK: Apparent Terminal Elimination Half-life (t1/2)
Description: Apparent terminal elimination half-life of LY3295668.
Time Frame: Cycle 1: Day 1 and Day 15: Predose, 1, 2, 4, 6, and 8-12 hours post-dose; Cycle 1: Day 2 and Day 8 Predose
Population: Zero participants analyzed due to data not collected.
Arm/Group | 25 mg LY3295668 (Phase 2)
Number analyzed (Participants) | 0

10. Secondary Outcome: Phase 2: PK: Apparent Total Plasma Clearance (CL/F)
Description: Apparent total plasma clearance of LY3295668.
Time Frame: Cycle 1: Day 1 and Day 15: Predose, 1, 2, 4, 6, and 8 -12 hours post-dose; Cycle 1: Day 2 and Day 8 Predose
Population: Zero participants analyzed due to data not collected.
Arm/Group | 25 mg LY3295668 (Phase 2)
Number analyzed (Participants) | 0

11. Secondary Outcome: Phase 2: PK: Apparent Volume of Distribution (Vz/F)
Description: Apparent volume of distribution of LY3295668.
Time Frame: Cycle 1: Day 1 and Day 15: Predose, 1, 2, 4, 6, and 8 -12 hours post-dose; Cycle 1: Day 2 and Day 8 Predose
Population: Zero participants analyzed due to data not collected.
Arm/Group | 25 mg LY3295668 (Phase 2)
Number analyzed (Participants) | 0

12. Secondary Outcome: Phase 1: Number of Participants With Worst Post-Baseline Grade >=3 White Blood Cell Count (WBC)
Description: Presented are participants with the worst post-baseline WBC Grade >= 3 using the National Cancer Institute (NCI) Common Terminology Criteria For Adverse Events version 4.03 (CTCAE v4.03). where Grade 1: < Lower Limit Normal (LLN) - 3000/mm3; <LLN - 3.0 x10e9/L, Grade 2: <3000 - 2000/mm3; <3.0 - 2.0 x10e9/L, Grade 3: <2000 - 1000/mm3; <2.0 1.0 x10e9/L, Grade 4: <1000/mm3; <1.0 x10e9/L.
Time Frame: Cycle 1 Day 1 through 30 Days After Treatment End Date (Up to 29 Months)
Population: All participants who received at least one dose of study drug, whether or not they completed all protocol requirements in Phase 1 per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg LY3295668 (Phase 1) | 50 mg LY3295668 (Phase 1) | 75 mg LY3295668 (Phase 1)
Number analyzed (Participants) | 8 | 2 | 2
Participants | 1 | 0 | 0

13. Secondary Outcome: Phase 1: Number of Participants With Worst Post-Baseline Grade >=3 Neutrophils (Segmented and Blended)
Description: Presented are participants with the worst post-baseline neutrophils Grade >=3 using the NCI-CTCAE v4.03 where Grade 1: < LLN - 1500/mm3; <LLN - 1.5 x10e9/L, Grade 2: <1500 - 1000/mm3; <1.5 - 1.0 x10e9/L, Grade 3: <1000 - 500/mm3; <1.0 - 0.5 x10e9/L, Grade 4: <500/mm3; <0.5 x 10e9/L.
Time Frame: Cycle 1 Day 1 through 30 Days After Treatment End Date (Up to 29 Months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg LY3295668 (Phase 1) | 50 mg LY3295668 (Phase 1) | 75 mg LY3295668 (Phase 1)
Number analyzed (Participants) | 8 | 2 | 2
Participants | 1 | 0 | 1

14. Secondary Outcome: Phase 1: Number of Participants With Worst Post-Baseline Grade >=3 Lymphocytes
Description: Presented are participants with the worst post-baseline lymphocytes Grade >=3 using the NCI-CTCAE version 4.03 where Grade 1: <LLN - <800/mm3, <LLN - 0.8 x 10e9/L, Grade 2: <800 - 500/mm3; <0.8 - 0.5 x 10e9/L, Grade 3: <500 - 200/mm3; <0.5 - 0.2 x 10e9/L, <200mm3; <0.2 x 10e9/L.
Time Frame: Cycle 1 Day 1 through 30 Days After Treatment End Date (Up to 29 Months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg LY3295668 (Phase 1) | 50 mg LY3295668 (Phase 1) | 75 mg LY3295668 (Phase 1)
Number analyzed (Participants) | 8 | 2 | 2
Participants | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 29 Months
Description: All participants who received at least one dose of study drug, whether or not they completed all protocol requirements. Gender specific events occurring only in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- 25 Milligrams (mg) LY3295668: 25 mg LY3295668 BID administered orally in 21-day cycles. Phase 1 and Phase 2 participants have been combined.
- 50 mg LY3295688: 50 mg LY3295668 BID administered orally in 21-day cycles.
- 75 mg LY3295688: 75 mg LY3295668 BID administered orally in 21-day cycles
Arm/Group | 25 Milligrams (mg) LY3295668 | 50 mg LY3295688 | 75 mg LY3295688
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 4/9 | 1/2 | 2/2
Other Adverse Events (participants affected / at risk) | 9/9 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 Milligrams (mg) LY3295668 (N=9) | 50 mg LY3295688 (N=2) | 75 mg LY3295688 (N=2)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Corneal deposits (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 25 Milligrams (mg) LY3295668 (N=9) | 50 mg LY3295688 (N=2) | 75 mg LY3295688 (N=2)
Anaemia (Blood and lymphatic system disorders) | 2 (34) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Night blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (4) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Gingival recession (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 5 (6) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 2 (4) | 2 (3)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parosmia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1/5 (1) | 0/1 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0/5 (0) | 0/1 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (5) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated due to sponsor decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/34/NCT03092934/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT03092934/SAP_001.pdf